CLINICAL TRIAL: NCT02214992
Title: Bioequivalence of 80 mg Telmisartan / 10 mg Ramipril Fixed Dose Combination Compared With the Monocomponents, Telmisartan and Ramipril (Two Different Formulations) Given Concomitantly to Healthy Male and Female Volunteers (an Open-label, Randomised, Single-dose, Three-way Crossover Study)
Brief Title: Bioequivalence of Telmisartan/g Ramipril Fixed Dose Combination Compared With the Monocomponents Telmisartan and Ramipril (Two Different Formulations) Given Concomitantly to Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1236.5
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Ramipril

ARMS (3):
- Telmisartan/Ramipril (Experimental): Fixed dose combination tablet
  Interventions: Drug: Telmisartan/Ramipril
- Telmisartan + Ramipril capsule (Active Comparator)
  Interventions: Drug: Telmisartan; Drug: Ramipril capsule
- Telmisartan + Ramipril tablet (Active Comparator)
  Interventions: Drug: Telmisartan; Drug: Ramipril tablet

INTERVENTIONS:
Drug: Telmisartan/Ramipril — Fixed dose combination tablet
  Arms: Telmisartan/Ramipril
Drug: Telmisartan
  Other Names: Micardis®
  Arms: Telmisartan + Ramipril capsule; Telmisartan + Ramipril tablet
Drug: Ramipril capsule
  Other Names: Altace®
  Arms: Telmisartan + Ramipril capsule
Drug: Ramipril tablet
  Other Names: Delix®
  Arms: Telmisartan + Ramipril tablet

SUMMARY:
Study to demonstrate the bioequivalence of 80 mg telmisartan/10 mg ramipril fixed dose combination versus its monocomponents given concurrently

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥ 18 and Age ≤ 55 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial (especially unspecific inducing agents like St.John´s wort (Hypericum perforatum) or inhibitors like cimetidine) or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during 24 hours prior to dosing and 24 hours after dosing
* Alcohol abuse (more than 60 g/day) or inability to stop alcoholic beverages for 24 hours prior to dosing and up to the last sampling time point, 96 hours after dosing
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hyperkalemia, hypokalemia, family history of Long QT Syndrome)
* Any history of relevant low blood pressure
* Supine blood pressure at screening of systolic <110 mm Hg and diastolic <60 mm Hg
* History of urticaria
* History of angioneurotic edema
* Hereditary fructose intolerance

For female subjects:

* Pregnancy or planning to become pregnant during the study or within 2 months of study completion
* Positive pregnancy test
* Are not willing or are unable to use a reliable method of contraception (such as implants, injectables and combined oral contraceptives, sterilisation, intrauterine device, double barrier method, sexual abstinence) for at least 1 month prior to participation in the trial, during and up to 1 month after completion/termination of the trial
* Chronic use of oral contraception or hormone replacement containing ethinyl estradiol as the only method of contraception
* Currently lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours after drug administration
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval from t1 to t2) | up to 96 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 96 hours after drug administration
λz (terminal rate constant in plasma) | up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 96 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | up to 96 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 96 hours after drug administration
Number of patients with adverse events | up to 78 days
Number of patients with clinically relevant changes in laboratory tests | up to 78 days
Number of patients with clinically relevant changes in Vital Signs (Blood Pressure, Pulse Rate) | up to 78 days
Number of patients with clinically relevant changes in 12-lead Electrocardiogram (ECG) | up to 78 days
Assessment of ttolerability by investigator on a 4-point scale | Day 5 of each treatment